CLINICAL TRIAL: NCT06714539
Title: Patient Specific Virtual Reality for Simulation of Spine Procedures: an Intelligent Image Segmentation, Registration and 3-dimensional Visualization in a Unified Virtual Reality Workflow for Image Guided Therapy, and Education - Physician Testing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Sunnybrook Research Institute (Other)
Responsible Party: Principal Investigator, Michael Hardisty, Scientist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 6489
Record Dates: First submitted 2024-11-25; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Surgical Education
Keywords: Surgical Education; Virtual Reality; Spine Surgery; Treatment Planning; Physician Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient Specific Virtual Reality Stimulation (Experimental): Physician participants will engage with the patient specific virtual reality simulator through multi-player teaching and individual practice modes.
  Interventions: Device: Patient Specific Virtual Reality Stimulation

INTERVENTIONS:
Device: Patient Specific Virtual Reality Stimulation — A novel virtual reality (VR) simulator for spine procedures that will take patient specific medical imaging (3D scans) and create a virtual patient that surgical procedures can be performed on.

SUMMARY:
The goal of this clinical trial is to learn if patient specific virtual reality (VR) simulations can be used for surgical orthopaedic education in resident and fellow physician populations.

DETAILED DESCRIPTION:
This project will combine advanced 3d visualization, interaction, medical image segmentation, and registration to create and integrate a virtual reality (VR) model into surgical orthopaedic education. The work has 3 aspects,

1) creating a patient specific 3D model with high accuracy of anatomic structures using patient specific medical imaging in an automated fashion, 2) interacting with 3D models of the patients, allowing the surgical procedures to be performed in virtual reality (including the resection of tissues, and placement of implants), 3) integrating the VR simulator into the surgical education of orthopaedic residents and fellows in training. This platform will reduce the time and cost associated with use of patient specific data, ultimately enabling pre-operative planning, post-procedural assessment and surgical simulation of spine procedures. The technology will improve surgical training, and the options for pre-treatment planning that will lead to better patient care, more efficient use of operating room time, and better trained surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Any resident of fellow physician enrolled in the participating site's spine surgery training program.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2024-12-02 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of patient specific VR surgical simulations for orthopaedic education, focusing on spinal decompression with or without instrumentation. | Up to 4 months for residents; up to 1 year for fellows
  Participants will complete study questionnaires before and after the testing sessions that ask them to list relevant structures involved in spinal decompression surgery. Participants will rate their confidence and motivation using the VR tool on a scale of 1 (highly confidence) to 10 (low confidence).

SECONDARY OUTCOMES:
Create a highly automated image analysis pipeline for the creation of patient specific 3D spine models with sufficient fidelity for surgical simulation. | Through study completion, an average of 5 years.
  The performance of the pipeline will be measured by the total registration error, quantifying overlap of segmentation of structures, and the distance between landmarks.
Perceived utility of high-fidelity simulation of surgical spine procedures that make use of patient specific models. | Through study completion, an average of 5 years.
  Orthopaedic residents and fellows will test the tool, following, they will fill out a questionnaire about the utility of the tool for learning and surgical planning. Participants will report their agreeableness to statements about the utility on a scale of 1 (strongly disagree) to 5 (strongly agree), and provide their own comments.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Michael Hardisty, Principal Investigator — Sunnybrook Research Institute

IPD SHARING:
Plan to Share IPD: Undecided
As a non-FDA regulated trial the investigators are unsure how useful the data will be externally, but will post if there is interest.

REFERENCES:
- [Background] Chen T, Zhang Y, Ding C, Ting K, Yoon S, Sahak H, Hope A, McLachlin S, Crawford E, Hardisty M, Larouche J, Finkelstein J. Virtual reality as a learning tool in spinal anatomy and surgical techniques. N Am Spine Soc J. 2021 Apr 14;6:100063. doi: 10.1016/j.xnsj.2021.100063. eCollection 2021 Jun. PMID 35141628